CLINICAL TRIAL: NCT04015310
Title: Quantitative Magnetic Resonance Imaging in Biliary Disease: Health Economics Study
Acronym: BISECT
Status: Withdrawn | Type: Observational
Why Stopped: Delays due to COVID prevented the start of recruitment and funding was no longer available.
Sponsor: Perspectum (Industry)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: EC-156
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Primary Sclerosing Cholangitis; PSC
Keywords: MRCP; MRCP+; PSC; Health economic
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- PSC patients attending outpatient: Primary sclerosing cholangitis, as defined by EASL and AASLD guidelines.
  Interventions: Device: Quantitative Multi parametric MRI and enhanced MRCP

INTERVENTIONS:
Device: Quantitative Multi parametric MRI and enhanced MRCP — Patients will have quantitative MRI and enhanced MRCP on addition to their standard of care

SUMMARY:
This is a health economic study on using quantitative magnetic resonance imaging in biliary disease. It is an observational study aiming to recruit 40 patients with Primary Sclerosing Cholangitis (PSC) in 12 months. The aim of the study is to assess the effect of result of enhanced Magnetic Resonance Cholangiopancreatography (MRCP+) on the physicians' diagnosis and/or plans for patients with suspected or confirmed PSC, compared with usual standard of care. This study also aims to identify the cost-effectiveness of adding MRCP+ to the standard care pathway.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC) is the greatest unmet need in modern liver medicine. There continue to be no direct bio-markers for the diagnosis and monitoring of biliary diseases such as PSC, constituting a major barrier to drug development and to poor patient outcomes. This project aims to validate an imaging platform, enhanced Magnetic Resonance Cholangiopancreatography, MRCP+, to improve the standard of care for patients by generating the real-world evidence needed to support clinical adoption.

Biliary diseases significantly increase the likelihood of developing sclerosing cholangitis (SC), causing major morbidity and mortality. Sclerosing cholangitis, a chronic inflammatory cholestatic condition, is exemplified by the primary idiopathic autoimmune condition PSC. In the absence of effective therapies, hindered by a lack of measurable trial endpoints (bio-markers), liver transplantation is the only life-extending intervention, with PSC accounting for 15% of all European liver transplantations. Furthermore, biliary complications occur in 5-32% of all liver transplantations. MRCP+ has the potential to significantly improve the outlook for patients.

At present, diagnosis requires cholangiopancreatography, either magnetic resonance (MRCP) or endoscopic retrograde (ERCP). The current standard ERCP is expensive, invasive, and associated with a high risk of morbidity. MRCP is less invasive and cheaper. However, both result in inconsistent qualitative interpretations. MRCP+ is the first device to enable direct quantitative measurement of biliary disease and addresses both European and US Liver society (EASL and AASLD) concerns that early changes of PSC are missed by MRCP, necessitating adequate visualisation and quantitative assessment.

MRCP+ both enhances MRCP images and yields advanced quantitative biliary measures. Initial experience shows significant clinical potential. This project will provide substantive evidence for clinical adoption via a real-world study including heath economics to evaluate the cost-effectiveness and impact on the clinical care pathway.

To achieve this, 40 patients were recruited from the University Hospitals Birmingham (UHB) who are attending the centre for either a review or diagnosis of PSC. The patients will follow their usual care pathway, being seen by the consultant who will document their care plan. Following this appointment, and their consent, they will be asked to undergo a non-invasive, pain-free Magnetic Resonance Imaging (MRI) scan. MRCP+ reports generated from these scans will be returned to the consultant who will review the documented standard care treatment plan and ascertain whether any amendments would have been made in light of these further quantitative metrics gained from MRI.

The study team alongside the Oxford Academic Health Science Network (OAHSN), will use the clinical data generated by the 40 patients and create a health economic model, which can be used to generate a business case for adoption, an impact case study for dissemination across the network of 15 centres in the Academic Health Science Networks (AHSN) and contribute to a submission for Human Tissue Authority (HTA) as part of the evidence required to gain health technology adoption via the National Institute for Health and Care Excellence (NICE) Medical Technologies Evaluation Programme (MTEP) route.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or over
* Patient due to attend the hepatology clinic for PSC diagnostics/review
* Participant is willing and able to give informed consent

Exclusion Criteria:

* The participants may not enter the study if they have any contraindication to magnetic resonance imaging (including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 adult participants will be recruited who are over the age of 18 and are attending a hepatology appointment at UHB and are either being investigated for PSC or have confirmed PSC.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
quantitative measurements using Enhance MRCP (MRCP+) and Physicians' decision making | 8 months
  To assess the effect of quantitative data from MRCP+ results on a physicians' diagnosis and/or plans for care of patients with suspected or confirmed PSC compared with usual standard of care.

SECONDARY OUTCOMES:
Cost effectiveness of using enhanced MRCP (MRCP+) for diagnosis and monitoring of PSC patients | 12 months
  To quantify the potential reduction in patient management costs by reducing unnecessary appointments in secondary care by using MRCP+ technology quantitative reports in diagnosis and monitoring of PSC patients more accurately.

IPD SHARING:
Plan to Share IPD: No